CLINICAL TRIAL: NCT03823456
Title: Self-acupressure for Cancer-related Symptom Cluster of Insomnia, Depression, and Anxiety in Cancer Patients: a Feasibility Randomized Controlled Trial
Brief Title: Self-acupressure for Cancer-related Symptom Cluster of Insomnia, Depression, and Anxiety: a Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20180604004
Record Dates: First submitted 2019-01-22; First posted 2019-01-30 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Insomnia; Anxiety; Depression
Keywords: acupressure; insomnia; anxiety; depression; symptom cluster
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression; Syndrome

STUDY DESIGN:
Intervention Model Description: True self-acupressure group [Enhanced standard care + True self-acupressure]:
  Participants will practice the four-week acupressure protocol plus standard care. During the four weeks treatment, participants will receive a weekly phone call follow up from researchers.
  Sham self-acupressure group [Enhanced standard care + Sham self-acupressure]:
  Patients will practice the four weeks sham self-acupressure protocol plus standard care. During the four weeks treatment, participants will receive a weekly follow up phone call from researchers.
  Enhanced standard care group The enhanced standard care in this study refers to standard care provided by the hospital includes health assessment, nutrition advice during taking chemotherapy treatment, hypnotics (Prescribe only where necessary by a doctor), and the enhanced care provided by the main researcher includes patient leaflet of tips on managing insomnia, depression, and anxiety; weekly follow-up phone call in four weeks.
Who Masked: Participant, Care Provider
Masking Description: In this study, due to the nature of the intervention, a partial double-blinded design will be employed. Participants randomize in standard care group will know their group assignment, but participants randomize to true and sham self-acupressure group will not know whether they receive true or sham self-acupressure treatment. Nevertheless, the outcomes of the study are all self-reported instruments, therefore, to some extent, the participants themselves could be viewed as "outcome assessors". Therefore, participants and "outcome assessors" located in true or sham self-acupressure group will be blinded on the treatment allocation. To ensure the successful blinding design, healthcare provider working in the wards will not know the group allocation, the main researcher will also work with the head-nurse of the department to arrange patient in intervention group and control groups into different wards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- True self-acupressure group (Experimental): True self-acupressure group [Enhanced standard care + True self-acupressure intervention protocol]:
  Participants in this group will practice the four-week acupressure protocol plus standard care. When participants admit hospital to receive chemotherapy treatment, they will receive a self-acupressure training section. Participants will be requested to practice acupressure at home once a day at night time (before going to bed) for four weeks. During the four weeks treatment, participants will receive a weekly phone call follow up from researchers.
  Interventions: Other: Self-acupressure
- Sham self-acupressure group (Placebo Comparator): Patients in this group will practice the four weeks sham self-acupressure protocol plus standard care. When participants admit hospital to receive chemotherapy treatment, they will receive a self-acupressure training section. Participants will be requested to practice sham acupressure at home once a day at night time (before going to bed) for four weeks. During the four weeks treatment, participants will receive a weekly follow up phone call from researchers
  Interventions: Other: Sham Self-acupressure
- Enhanced standard care group (No Intervention): The standard care for cancer patients undergoing chemotherapy includes health assessment, regular health advice regarding symptoms that patients report and nutrition advice during taking chemotherapy treatment. Apart from the standard care, we provide participants a leaflet with 10 recommendations which help participants manage insomnia, depression, and anxiety. By providing this leaflet, we slightly enhance the standard care but do not contaminate the effective of the intervention since these tips are basic and participants can easily read about them on the internet or newspaper. In addition, to minimize the bias caused by contacting between interventionist and participants, we also provide participants in the enhanced standard care group weekly follow up phone call in four weeks.

INTERVENTIONS:
Other: Self-acupressure — We teach participants how to using self-acupressure to manage insomnia, depression, and anxiety. Six acupoints are included in our acupressure protocol which are Baihui, Yintang, Fengchi, Neiguan, Shenmen, and Taichong. Participants are requested to stimulate each acupoint in 3 minutes once a day (at night time before going to bed) in 28 days (4 weeks). During the four weeks treatment, participants will receive a weekly phone call follow up to remind them practice self-acupressure at home. Participant also receives a patient leaflet with 10 tips heil to manage insomnia, depression, and anxiety. These tips include some basic sleep hygiene rules and tips to manage anxiety and depression adapted from Anxiety and Depression Association of American.
  Arms: True self-acupressure group
Other: Sham Self-acupressure — We using a sham acupressure protocol to teach participants in this group. Six sham acupoints are included in the protocol. The sham acupoints are located 2-5cm away from the true acupoints. Participants are requested to stimulate each sham acupoint in 3 minutes once a day (at night time before going to bed) in 28 days (4 weeks). During the four weeks treatment, participants will receive a weekly phone call follow up to remind them practice self-acupressure at home. Participant also receives a patient leaflet with 10 tips heil to manage insomnia, depression, and anxiety. These tips include some basic sleep hygiene rules and tips to manage anxiety and depression adapted from the Anxiety and Depression Association of American.
  Arms: Sham self-acupressure group

SUMMARY:
Aim: To assess the acceptability and make estimations about the effectiveness of using self-acupressure to manage insomnia, depression, and anxiety in cancer patients undergoing chemotherapy.

Study design: three-arms randomized sham-controlled trial. Participants will be assigned to the true self-acupressure group, sham acupressure group, or enhanced standard care group, with a ratio of 1:1:1 using block randomize.

Participants: patients receiving chemotherapy. 114 patients will be recruited to the study.

Inclusion criteria: Undergoing chemotherapy currently, Age 20 - 84 years' old, able to read and write Vietnamese, Karnofsky score ≥ 80, Insomnia Severity Index (ISI) score ≥ 11, Anxiety score measured by The Hospital Anxiety and Depression Scale (HADS) ≥ 8 and Depression score measured by HADS ≥ 8

Exclusion criteria:

Patients are excluded from the trial if they are unable to understand or cooperate with study procedures, receiving other cancer treatments (e.g., radiotherapy, hormonal therapy) at the same time as receiving chemotherapy and during the period of their involvement in the trial, participating in other research studies which may have interacted with the current trial or affect insomnia, depression, anxiety perception, having difficulties or are unable to practice self-acupressure by themselves, are receiving insomnia or depression/anxiety treatment currently.

Interventions Self-administered acupressure training section Participants in the true or sham self-acupressure groups will receive a self-administered acupressure training section based on their group assignment. Then, they will be requested to practice acupressure at home for 4 weeks.

Patient leaflet All of the participants in three groups will receive a patient leaflet with tips to manage insomnia, depression, and anxiety.

Weekly telephone reminder will be made to follow-up participants in all groups. Outcome measurement The recruitment rate, consent rate, refusal rate, attrition rate, adherence rate will be calculated. The acceptability of the intervention will be measured by the Intervention Rating Profile - 15. The ISI, The HADS, and The Functional Assessment of Cancer Therapy-General will be used to evaluate the effects of self-acupressure on the severity of insomnia, depression, anxiety. Others sleep parameters and adverse events associated with self-acupressure will be recorded.

DETAILED DESCRIPTION:
1. Background Major treatments for cancer include surgery, radiotherapy, and chemotherapy improve patient's survival but also can exert a significant psychosocial and physical impact on patients by producing a variety of unpleasant symptoms. Applying the concept of identification symptom cluster by the correlation between symptoms, different sleep-related symptom clusters among cancer patient have been identified across studies such as: fatigue, depression and insomnia; pain, fatigue and or pain, depression, and insomnia. However, the correlation between insomnia and other symptoms was not fully explored. Therefore, to identify current evidence of sleep-related symptom cluster, we have conducted a cross-sectional survey among 213 cancer patients undergoing chemotherapy in Vietnam. The results indicated that among participants, a symptom cluster of insomnia, depression, and anxiety was evident.

   Based on the literature review, acupressure can potentially reduce insomnia as well as other symptoms in cancer patients. However, the use of acupressure in specific self-acupressure in managing symptom cluster of insomnia, depression, and anxiety is unknown but worthy for further research.
2. Methodologies of the study 2.1. The development of the self-acupressure protocols for managing insomnia, depression, and anxiety To distinguish the specific treatment (true) effects of acupressure treatment from the nonspecific treatment (placebo) effects, a true self-acupressure protocol and a sham self-acupressure protocol were being developed accordingly. The true acupressure protocol was developed based on the theory of Traditional Chinese Medicine (TCM), available systematic reviews are used for selecting acupoints and choosing treatment dose, and World Health Organization (WHO) standard acupuncture point location guidelines were used to locate the acupoint and technique for self-acupressure.

True and sham acupressure protocol These acupoints are being selected for the true acupressure protocol Baihui (GV20), Yintang (EX-HN3), Fengchi (GB20), Neiguan (PC6), Shenmen (HT7), Taichong (LR3) These points are being selected for the sham acupressure protocol SA 1: Base of metacarpal bone of the right middle finger SA 2 2 cm superior to the end of the right eyebrow SA 3 Mastoid bone SA 4 Head of ulnar styloid SA 5 Base of metacarpal bone of the index finger SA 6 Medial malleolus Duration of each section (true and sham acupressure): 24 minutes (3 mins per point) Duration of whole treatment (true and sham acupressure): 4 weeks (28 days) Time for practice self-acupressure: Before bedtime (final activities of the day, after practicing acupressure the participants should attempt to sleep) The suitability of true and sham self-acupressure protocols had been validated by a panel of six TCM experts from Hong Kong and Vietnam.

2.2. Methods of the feasibility study 2.2.1. The study design A feasibility study with three-arms randomized sham-controlled trial will be set up. The three arms are the true acupressure group, the sham acupressure group, and the enhanced standard care group.

2.2.2. Sample size Applying the rule of thumb, 30 subjects will be recruited for each study groups. The potential drop-out rate of 20% is used to calculate the total sample size for the feasibility study. Therefore, the sample size will be set at 114 patients with 38 patients per group.

2.2.3. Settings The study will be conducted in the Vietnam National Cancer Institute and Hanoi Oncology Hospital. All of them are located in Hanoi, the capital of Vietnam.

2.2.4. Randomization, allocation concealment, and blinding 2.2.4.1. Randomization and allocation concealment. Block randomization will be. 114 participants will be randomized into three study groups in a block of six participants. A randomization table will be computer generated by using the online randomizer. It will be prepared and kept by a researcher who does not involve in any research process. After recruiting enough participants for a block, the main researcher will send the list of participants' name to the randomization table keeper. The randomization table keeper will then randomly assign participants into trial groups based on the prepared randomization table and email the group assignments to the main researcher.

2.2.4.2. Blinding Participants randomized in the standard care group will know their group assignment, but participants randomize to the true and sham self-acupressure group will not know whether they receive true or sham self-acupressure treatment. Nevertheless, the outcomes of the study are all self-reported instruments, so the participants themselves could be viewed as "outcome assessors". Therefore, participants and "outcome assessors" located in the true or sham self-acupressure group will be blinded on the treatment allocation.

2.2.5. Study procedures Participants from five chemotherapy units will be recruited to the study (two chemotherapy units in hospital A, and three from hospital B). On the first day patients admitted to the hospital, during the health assessment, nurses will ask the patients to rate the severity of insomnia, depression and anxiety that they experience during the previous month. Each of the symptoms will be measured by separate Numerical Analog Scales (NAS). NAS is an 11-point scales with 0 means "not present" and 10 means "worst possible". If the patients rate 4 or above for their insomnia, depression, and anxiety nurses will inform the main researcher and introduce the potential patient to the main researcher. The main researcher will introduce the study in detail to potential participants and give them the information sheet and inform consent form. After signing the consent form, researchers will collect the demographic data of participants and instruct participants to complete the baseline assessment. After the participants complete the baseline assessment, the main researcher will summarize the result and if the participants eligible for the trial they will be instructed how to complete the seven days sleep diary after they discharge from the hospital. Afterward, participants will be randomly assigned to one of the following groups: the true self-acupressure group (TSA), the sham self-acupressure group (SSA) and enhanced standard care group (ESC).

Participants in the true self-acupressure group or sham self-acupressure group Participants in these group will either receive a true self-acupressure or sham acupressure training section based on their group assignment. Participants will be requested to practice acupressure at home for four weeks after they complete the sleep diary baseline assessment (a telephone reminder will be made). During the four weeks treatment, participants will receive a weekly phone call from researchers for encouraging to practice acupressure and answer inquiries may have. During this period, participant will be requested to complete Self-acupressure record form every day. After four weeks treatment, participants will be asked to complete and send back all the post-intervention assessing questionnaire to research by express service. A short-term follow up will be then carried out in four weeks to assess the persistence effect of acupressure on the symptoms outcome. During this time, the patient will not practice acupressure at home. By the end of follow up time, researchers will make a telephone reminder to participants and ask them to complete and send back all the follow-up assessment questionnaire to the main research by express service. 200,000 Vietnam dong (vnd) will be given to participants for the express service charge by the end of the follow-up time.

Participants in the enhanced standard control group Participants in the enhanced standard control group will receive the leaflet with tips to manage insomnia, depression, and anxiety. Weekly telephone reminder will also be made in four weeks. By the end of week fourth, participants in this group will be requested to complete post-intervention assessment and send back to research by post. A short-term follow up will be then carried out in 4 weeks. During the follow-up period, participants receive no weekly telephone reminder. By the end of follow up time, researchers will make a telephone reminder to participants and ask them to complete and send back all the follow-up assessment questionnaire to research by express service. 200,000 vnd will be given to participants for the express service charge by the end of the follow-up time.

2.2.5.1. Training of Subject recruitment Five nurses will be recruited for subject recruitment. Nurses who work in potential chemotherapy units with at least one year of experience in working with cancer patients will be recruited. They will receive a training section conducted by the main researcher on how to recruite participants.

2.2.5.2. Training of the interventionists Four nurses will be trained to become interventionists for the study (2 nurses/hospital). Nurses who work in potential hospitals with at least two years of experience in working with cancer patients will be recruited as interventionists of the study. A one hours training section (TOT section) will be delivered by the main researcher and a TCM professional.

2.2.5.3. Training of the participants in the true self-acupressure group and sham self-acupressure group: Participants locate in these groups will receive education section. The training will be conducted in a group of two to four participants in 45 minutes. The self-acupressure training section will take place in the consultation room in the chemotherapy unit. In the education section, interventionists will instruct the participants how to locate and stimulate acupoint following the acupressure protocols. After giving instruction and time for participants to practice, interventionists checksthe patient's mastery of self-acupressure technique by using the Acupressure Skill Check form for participants. If the participant fails to identify the acupoint or stimulate the acupoint wrongly, the interventionist will then correct them. By the end of the education section, a patient booklet includes step by step guideline with images-illustrating acupressure protocol will be given to participants.

2.3. Ethical consideration The study had gained ethical approval from The Hong Kong Polytechnic University and Vietnamese Ministry of Health. This study has followed the ethical principles for research that involves human subjects which are: autonomy, beneficence, non-maleficence, and confidentiality).

2.4. Data Analysis Data will be checked for normality, outliers, and missing data. Intention to treat principle is adapted for analyzing the result of the pilot study which use the "last value carried out forward" approach to replace missing data. Descriptive statistics will be used to analyze the sample characteristics, demographics, and data related to the intervention feasibility, acceptability and adverse event of acupressure. Baseline differences among the three groups will be compared by chi-square test and repeated measure ANOVA. In case the chi-square test is not appropriated because of low cell counts (≤ 5), it will be replaced by Fisher's exact test. The effect size will be calculated by Cohen d based on the mean difference between baseline and end of the treatment period for each symptom and the cluster of insomnia, depression, and anxiety in the true self-acupressure group and sham acupressure group. The significance level is set at 0.05. IBM SPSS 20.0 software will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing chemotherapy currently.
* Able to read and write Vietnamese (to complete the questionnaires and provide informed consent).
* Have Karnofsky score ≥ 80 (to be able to practice self-acupressure).
* Have Insomnia Severity Index score ≥ 11
* Have Anxiety score measured by HADS ≥ 8 and Depression score measured by HADS ≥ 8

Exclusion Criteria:

* Are unable to understand or cooperate with study procedures.
* Are receiving other cancer treatments (e.g., radiotherapy, hormonal therapy) at the same time as receiving chemotherapy and during the period of their involvement in the trial.
* Are participating in other research studies which may have interacted with the current trial or affect insomnia, depression, anxiety perception.
* Have difficulties or are unable to practice self-acupressure by themselves.
* Are receiving insomnia or depression/anxiety treatment currently.

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of eligible participants | up to 15 weeks
  The recruitment rate is calculated by dividing the number of the eligible participant by the total number of screened participants
Number of patients who refuse to participant in the study | up to 15 weeks
  The refusal rate is calculated by dividing the number of participants who do not participate in the study by the total number of eligible participants
Acceptability score of the intervention measured by participants | One month after participants enroll the trial
  The acceptability score of the intervention will be measured by The Intervention Rating Profile - 15 (Martens, Witt, Elliott, & Darveaux, 1985). The Intervention Rating Profile - 15 (IRP-15) consists of 15 items; each item is rated on a six-point Likert scale ranging from one (Strongly disagree) to six (Strongly agree). The higher score indicated higher acceptability of the intervention. The scale had been validated, translated into Vietnamese with high reliability (Cronbach's α = 0.89) (Nguyen, Alexander, & Yates, 2018)
Acceptability of study procedures measured by participants | One month after participants enroll the trial
  The attrition rate will be calculated by the number of participants who decide to discontinue the study and the number of participants who are lost to contact during the study period. Reason for dropping out and lost to contact will be recorded
Adverse events associated with self-acupressure reported by participants | One month after participants enroll the trial
  Participants will be requested to report potential adverse events related to acupressure in the "Self-Acupressure Record Form."
Change from baseline in insomnia score on Insomnia Severity Index at post intevention and after follow-up time | Change from baseline insomnia severity at one month and two months
  The Insomnia Severity Index (ISI) is used to measure insomnia severity among participants. The ISI is a self-reported questionnaire consisting of seven items to assess the nature, severity, and impact of insomnia. A score of 7 items indicates the insomnia severity, the min score is 0 and the maximum score is 28, the higher score indicates worse insomnia severity. The insomnia severity is interpreted as follows: moderate insomnia (ISI score of 15 to 21), severe insomnia (ISI score of 22 to 28). This instrument had been validated translated into Vietnamese previously (Long, Thanasilp, & Thato, 2016) and was being used in our previous study with high reliability (Cronbach's α = 0.92).
Change of participants' sleep parameter in sleep diary from baseline at post intervention and after follow-up time | Change from baseline at one month and two months
  A sleep diary is used to measure sleep parameters. The participant will be requested to complete a one-week sleep diary before starting practice acupressure, after the treatment period ends, and after. The sleep diary is used to measure these sleep parameters: Total Sleep time (minute), total time in bed (minute), the number of night awaken after sleep onset and sleep efficiency.
Change from baseline in depression and anxiety scoreon Hospital Depression and Anxiety Scale at post intevention and after follow-up time | Change from baseline depression and anxiety severity at one month and two months
  The Hospital Anxiety and Depression Scale (HADS) was developed by Zigmond and Snaith (1983) to measure depression and anxiety among participants. This scale has 14 items, seven items measuring anxiety and seven items measuring depression over the past week. The total depression/anxiety score range from 0 to 28 with the higher total score indicates worse depression/anxiety. This instrument had been translated into Vietnamese previously (Long et al., 2016) and was used in our previous study with the Cronbach's alpha for the scale was 0.87, and for anxiety, subscale was 0.86, and for depression, subscale was 0.76.
Change from baseline in symptom cluster score on numerical analo scale from baseline at post intervetion and after follow-up time | Change from baseline symptom cluster severity at one month and two months
  Separate numerical analog scales (NAS) for each symptom will be used to measure the severity of the whole cluster in the previous month. The symptom severity score of each of symptom in the cluster will be measured by an 11-point scales with 0 means "not present" and 10 means "as bad as it could be." Symptom severity at the cluster level will be evaluated by the averaging symptom severity score of each symptom in the cluster.
Change in participants'quality of life on the Functional Assessment of Cancer Therapy-General scale from baseline at post intervention and after follow-up time | Change from baseline quality of life at one month and two months
  The Functional Assessment of Cancer Therapy-General (FACT-G) is used in this study to assess the quality of life in participants. The questionnaire consists of 27 items each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). This scale measures four sub-scales: Physical well-being (PWB, 7 items); Social/family well-being (SWB, 7 items); Emotional well-being (EWB, 6 items) and Functional well-being (FWB, 7 items). The total score range from 0 to 108, questions are phrased so that higher numbers indicate a better health state. Each subscale is scored, and a total score for the FACT-G is obtained by adding each of the subscale scores. This instrument has been translated into Vietnamese by the Functional Assessment of Chronic Illness Therapy system and had been used in the previous study with the Cronbach's alpha for the scale was 0.89, and for Emotional well-being, subscales were 0.78, FWB = 0.82, PWB = 0.81 and for SWB was 0.82.

CONTACTS AND LOCATIONS:
Overall Officials: Huong TX Hoang, Study Director — The Hong Kong Polytechnic University; Alex Molassiotis, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Vietnam (2):
  - Vietnam National Cancer Institution, Hanoi, Ha Dong
  - Hanoi Oncology Hospital, Hanoi, Hai Ba Trung

IPD SHARING:
Plan to Share IPD: No
As required by ethical principals, we will not share IPD to other researchers in order to protect the participant's personal information.

REFERENCES:
- [Background] Abedian Z, Eskandari L, Abdi H, Ebrahimzadeh S. The Effect of Acupressure on Sleep Quality in Menopausal Women: A Randomized Control Trial. Iran J Med Sci. 2015 Jul;40(4):328-34. PMID 26170519
- [Background] Altman DG, Schulz KF, Moher D, Egger M, Davidoff F, Elbourne D, Gotzsche PC, Lang T; CONSORT GROUP (Consolidated Standards of Reporting Trials). The revised CONSORT statement for reporting randomized trials: explanation and elaboration. Ann Intern Med. 2001 Apr 17;134(8):663-94. doi: 10.7326/0003-4819-134-8-200104170-00012. PMID 11304107
- [Background] Anderson KO, Getto CJ, Mendoza TR, Palmer SN, Wang XS, Reyes-Gibby CC, Cleeland CS. Fatigue and sleep disturbance in patients with cancer, patients with clinical depression, and community-dwelling adults. J Pain Symptom Manage. 2003 Apr;25(4):307-18. doi: 10.1016/s0885-3924(02)00682-6. PMID 12691682
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Bokmand S, Flyger H. Acupuncture relieves menopausal discomfort in breast cancer patients: a prospective, double blinded, randomized study. Breast. 2013 Jun;22(3):320-3. doi: 10.1016/j.breast.2012.07.015. Epub 2012 Aug 18. PMID 22906948
- [Background] Bonnet MH, Arand DL. Sleepiness as measured by modified multiple sleep latency testing varies as a function of preceding activity. Sleep. 1998 Aug 1;21(5):477-83. PMID 9703587
- [Background] Buysse DJ, Ancoli-Israel S, Edinger JD, Lichstein KL, Morin CM. Recommendations for a standard research assessment of insomnia. Sleep. 2006 Sep;29(9):1155-73. doi: 10.1093/sleep/29.9.1155. PMID 17040003
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Cerrone R, Giani L, Galbiati B, Messina G, Casiraghi M, Proserpio E, Meregalli M, Trabattoni P, Lissoni P, Gardani G. Efficacy of HT 7 point acupressure stimulation in the treatment of insomnia in cancer patients and in patients suffering from disorders other than cancer. Minerva Med. 2008 Dec;99(6):535-7. PMID 19034252
- [Background] Choi TY, Kim JI, Lim HJ, Lee MS. Acupuncture for Managing Cancer-Related Insomnia: A Systematic Review of Randomized Clinical Trials. Integr Cancer Ther. 2017 Jun;16(2):135-146. doi: 10.1177/1534735416664172. Epub 2016 Aug 16. PMID 27531549
- [Background] Chung KF, Yeung WF, Yu YM, Yung KP, Zhang SP, Zhang ZJ, Wong MT, Lee WK, Chan LW. Acupuncture for residual insomnia associated with major depressive disorder: a placebo- and sham-controlled, subject- and assessor-blind, randomized trial. J Clin Psychiatry. 2015 Jun;76(6):e752-60. doi: 10.4088/JCP.14m09124. PMID 26132682
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Freemantle N, Calvert M, Wood J, Eastaugh J, Griffin C. Composite outcomes in randomized trials: greater precision but with greater uncertainty? JAMA. 2003 May 21;289(19):2554-9. doi: 10.1001/jama.289.19.2554. PMID 12759327
- [Background] Dowrick AS, Bhandari M. Ethical issues in the design of randomized trials: to sham or not to sham. J Bone Joint Surg Am. 2012 Jul 18;94 Suppl 1:7-10. doi: 10.2106/JBJS.L.00298. PMID 22810439
- [Background] Grady C. Payment of clinical research subjects. J Clin Invest. 2005 Jul;115(7):1681-7. doi: 10.1172/JCI25694. PMID 16007244
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Hollis S, Campbell F. What is meant by intention to treat analysis? Survey of published randomised controlled trials. BMJ. 1999 Sep 11;319(7211):670-4. doi: 10.1136/bmj.319.7211.670. PMID 10480822
- [Background] Hrobjartsson A, Gotzsche PC. Placebo interventions for all clinical conditions. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD003974. doi: 10.1002/14651858.CD003974.pub3. PMID 20091554
- [Background] Hughes JG, Russell W, Breckons M, Richardson J, Lloyd-Williams M, Molassiotis A. "I assumed that one was a placebo": exploring the consent process in a sham controlled acupressure trial. Complement Ther Med. 2014 Oct;22(5):903-8. doi: 10.1016/j.ctim.2014.07.005. Epub 2014 Jul 19. PMID 25440382
- [Background] Juni P, Altman DG, Egger M. Systematic reviews in health care: Assessing the quality of controlled clinical trials. BMJ. 2001 Jul 7;323(7303):42-6. doi: 10.1136/bmj.323.7303.42. No abstract available. PMID 11440947
- [Background] Kwekkeboom KL. Cancer Symptom Cluster Management. Semin Oncol Nurs. 2016 Nov;32(4):373-382. doi: 10.1016/j.soncn.2016.08.004. Epub 2016 Oct 24. PMID 27789073
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Landolt HP, Roth C, Dijk DJ, Borbely AA. Late-afternoon ethanol intake affects nocturnal sleep and the sleep EEG in middle-aged men. J Clin Psychopharmacol. 1996 Dec;16(6):428-36. doi: 10.1097/00004714-199612000-00004. PMID 8959467
- [Background] Lee EJ, Frazier SK. The efficacy of acupressure for symptom management: a systematic review. J Pain Symptom Manage. 2011 Oct;42(4):589-603. doi: 10.1016/j.jpainsymman.2011.01.007. Epub 2011 Apr 30. PMID 21531533
- [Background] Levine RJ. What should consent forms say about cash payments? IRB. 1979 Oct;1(6):7-8. No abstract available. PMID 11661756
- [Background] Lu MJ, Lin ST, Chen KM, Tsang HY, Su SF. Acupressure improves sleep quality of psychogeriatric inpatients. Nurs Res. 2013 Mar-Apr;62(2):130-7. doi: 10.1097/NNR.0b013e3182781524. PMID 23302821
- [Background] Lynn MR. Determination and quantification of content validity. Nurs Res. 1986 Nov-Dec;35(6):382-5. No abstract available. PMID 3640358
- [Background] Mao JJ, Bowman MA, Xie SX, Bruner D, DeMichele A, Farrar JT. Electroacupuncture Versus Gabapentin for Hot Flashes Among Breast Cancer Survivors: A Randomized Placebo-Controlled Trial. J Clin Oncol. 2015 Nov 1;33(31):3615-20. doi: 10.1200/JCO.2015.60.9412. Epub 2015 Aug 24. PMID 26304905
- [Background] Murphy SL, Gutman SA. Intervention fidelity: a necessary aspect of intervention effectiveness studies. Am J Occup Ther. 2012 Jul-Aug;66(4):387-8. doi: 10.5014/ajot.2010.005405. No abstract available. PMID 22742685
- [Background] Nehlig A. Are we dependent upon coffee and caffeine? A review on human and animal data. Neurosci Biobehav Rev. 1999 Mar;23(4):563-76. doi: 10.1016/s0149-7634(98)00050-5. PMID 10073894
- [Background] Nguyen LT, Alexander K, Yates P. Psychoeducational Intervention for Symptom Management of Fatigue, Pain, and Sleep Disturbance Cluster Among Cancer Patients: A Pilot Quasi-Experimental Study. J Pain Symptom Manage. 2018 Jun;55(6):1459-1472. doi: 10.1016/j.jpainsymman.2018.02.019. Epub 2018 Mar 2. PMID 29505795
- [Background] Paterson C, Dieppe P. Characteristic and incidental (placebo) effects in complex interventions such as acupuncture. BMJ. 2005 May 21;330(7501):1202-5. doi: 10.1136/bmj.330.7501.1202. PMID 15905259
- [Background] Pilkington K. Anxiety, depression and acupuncture: A review of the clinical research. Auton Neurosci. 2010 Oct 28;157(1-2):91-5. doi: 10.1016/j.autneu.2010.04.002. Epub 2010 May 6. PMID 20451469
- [Background] Pilkington K, Kirkwood G, Rampes H, Cummings M, Richardson J. Acupuncture for anxiety and anxiety disorders--a systematic literature review. Acupunct Med. 2007 Jun;25(1-2):1-10. doi: 10.1136/aim.25.1-2.1. PMID 17641561
- [Background] Probst P, Grummich K, Heger P, Zaschke S, Knebel P, Ulrich A, Buchler MW, Diener MK. Blinding in randomized controlled trials in general and abdominal surgery: protocol for a systematic review and empirical study. Syst Rev. 2016 Mar 24;5:48. doi: 10.1186/s13643-016-0226-4. PMID 27012940
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Sok SR, Erlen JA, Kim KB. Effects of acupuncture therapy on insomnia. J Adv Nurs. 2003 Nov;44(4):375-84. doi: 10.1046/j.0309-2402.2003.02816.x. PMID 14651709
- [Background] Song HJ, Seo HJ, Lee H, Son H, Choi SM, Lee S. Effect of self-acupressure for symptom management: a systematic review. Complement Ther Med. 2015 Feb;23(1):68-78. doi: 10.1016/j.ctim.2014.11.002. Epub 2014 Dec 4. PMID 25637155
- [Background] Spence DW, Kayumov L, Chen A, Lowe A, Jain U, Katzman MA, Shen J, Perelman B, Shapiro CM. Acupuncture increases nocturnal melatonin secretion and reduces insomnia and anxiety: a preliminary report. J Neuropsychiatry Clin Neurosci. 2004 Winter;16(1):19-28. doi: 10.1176/jnp.16.1.19. PMID 14990755
- [Background] Sun JL, Sung MS, Huang MY, Cheng GC, Lin CC. Effectiveness of acupressure for residents of long-term care facilities with insomnia: a randomized controlled trial. Int J Nurs Stud. 2010 Jul;47(7):798-805. doi: 10.1016/j.ijnurstu.2009.12.003. Epub 2010 Jan 6. PMID 20056221
- [Background] Tan JY, Suen LK, Wang T, Molassiotis A. Sham Acupressure Controls Used in Randomized Controlled Trials: A Systematic Review and Critique. PLoS One. 2015 Jul 15;10(7):e0132989. doi: 10.1371/journal.pone.0132989. eCollection 2015. PMID 26177378
- [Background] Tickle-Degnen L. Nuts and bolts of conducting feasibility studies. Am J Occup Ther. 2013 Mar-Apr;67(2):171-6. doi: 10.5014/ajot.2013.006270. PMID 23433271
- [Background] Tough EA, White AR, Richards SH, Lord B, Campbell JL. Developing and validating a sham acupuncture needle. Acupunct Med. 2009 Sep;27(3):118-22. doi: 10.1136/aim.2009.000737. PMID 19734382
- [Background] Tsay SL, Chen ML. Acupressure and quality of sleep in patients with end-stage renal disease--a randomized controlled trial. Int J Nurs Stud. 2003 Jan;40(1):1-7. doi: 10.1016/s0020-7489(02)00019-6. PMID 12550145
- [Background] Vickers AJ. How to randomize. J Soc Integr Oncol. 2006 Fall;4(4):194-8. doi: 10.2310/7200.2006.023. PMID 17022927
- [Background] Viera AJ, Bangdiwala SI. Eliminating bias in randomized controlled trials: importance of allocation concealment and masking. Fam Med. 2007 Feb;39(2):132-7. PMID 17273956
- [Background] Waits A, Tang YR, Cheng HM, Tai CJ, Chien LY. Acupressure effect on sleep quality: A systematic review and meta-analysis. Sleep Med Rev. 2018 Feb;37:24-34. doi: 10.1016/j.smrv.2016.12.004. Epub 2016 Dec 22. PMID 28089414
- [Background] Wang H, Qi H, Wang BS, Cui YY, Zhu L, Rong ZX, Chen HZ. Is acupuncture beneficial in depression: a meta-analysis of 8 randomized controlled trials? J Affect Disord. 2008 Dec;111(2-3):125-34. doi: 10.1016/j.jad.2008.04.020. Epub 2008 Jun 11. PMID 18550177
- [Background] Werth E, Dijk DJ, Achermann P, Borbely AA. Dynamics of the sleep EEG after an early evening nap: experimental data and simulations. Am J Physiol. 1996 Sep;271(3 Pt 2):R501-10. doi: 10.1152/ajpregu.1996.271.3.R501. PMID 8853369
- [Background] Wetter DW, Fiore MC, Baker TB, Young TB. Tobacco withdrawal and nicotine replacement influence objective measures of sleep. J Consult Clin Psychol. 1995 Aug;63(4):658-67. doi: 10.1037//0022-006x.63.4.658. PMID 7673544
- [Background] Williams JM, Kay DB, Rowe M, McCrae CS. Sleep discrepancy, sleep complaint, and poor sleep among older adults. J Gerontol B Psychol Sci Soc Sci. 2013 Sep;68(5):712-20. doi: 10.1093/geronb/gbt030. Epub 2013 Jun 26. PMID 23804432
- [Background] Xiang Y, He JY, Li R. Appropriateness of sham or placebo acupuncture for randomized controlled trials of acupuncture for nonspecific low back pain: a systematic review and meta-analysis. J Pain Res. 2017 Dec 28;11:83-94. doi: 10.2147/JPR.S152743. eCollection 2018. PMID 29343984
- [Background] World Health Organization. (2009). WHO Standard Acupuncture point locations in the Western Pacific Region.
- [Background] World Medical Association Inc. Declaration of Helsinki. Ethical principles for medical research involving human subjects. J Indian Med Assoc. 2009 Jun;107(6):403-5. No abstract available. PMID 19886379
- [Background] Yang XY, Shi GX, Li QQ, Zhang ZH, Xu Q, Liu CZ. Characterization of deqi sensation and acupuncture effect. Evid Based Complement Alternat Med. 2013;2013:319734. doi: 10.1155/2013/319734. Epub 2013 Jun 20. PMID 23864884
- [Background] Yeung WF, Chung KF, Poon MM, Ho FY, Zhang SP, Zhang ZJ, Ziea ET, Wong VT. Acupressure, reflexology, and auricular acupressure for insomnia: a systematic review of randomized controlled trials. Sleep Med. 2012 Sep;13(8):971-84. doi: 10.1016/j.sleep.2012.06.003. Epub 2012 Jul 25. PMID 22841034
- [Background] Yeung WF, Chung KF, Poon MM, Ho FY, Zhang SP, Zhang ZJ, Ziea ET, Wong Taam V. Prescription of chinese herbal medicine and selection of acupoints in pattern-based traditional chinese medicine treatment for insomnia: a systematic review. Evid Based Complement Alternat Med. 2012;2012:902578. doi: 10.1155/2012/902578. Epub 2012 Nov 28. PMID 23259001
- [Background] Yeung WF, Ho FY, Chung KF, Zhang ZJ, Yu BY, Suen LK, Chan LY, Chen HY, Ho LM, Lao LX. Self-administered acupressure for insomnia disorder: a pilot randomized controlled trial. J Sleep Res. 2018 Apr;27(2):220-231. doi: 10.1111/jsr.12597. Epub 2017 Sep 8. PMID 28884877
- [Background] Young, J. S. (2001). Acupressure : simple steps to health : discover your body's powerpoints for health and relaxation ([New ed.]. ed.). London: London : Thorsons.
- [Background] Zhang H, Bian Z, Lin Z. Are acupoints specific for diseases? A systematic review of the randomized controlled trials with sham acupuncture controls. Chin Med. 2010 Jan 12;5:1. doi: 10.1186/1749-8546-5-1. PMID 20145733
- [Background] Zheng, L.-W., Chen, Y., Chen, F., Zhang, P., & Wu, L.-F. (2014). Effect of acupressure on sleep quality of middle-aged and elderly patients with hypertension (Vol. 1).
- [Background] Zick SM, Sen A, Wyatt GK, Murphy SL, Arnedt JT, Harris RE. Investigation of 2 Types of Self-administered Acupressure for Persistent Cancer-Related Fatigue in Breast Cancer Survivors: A Randomized Clinical Trial. JAMA Oncol. 2016 Nov 1;2(11):1470-1476. doi: 10.1001/jamaoncol.2016.1867. PMID 27388752
- [Derived] Hoang HTX, Molassiotis A, Chan CW, Vu AH, Bui PT. Pilot randomized sham-controlled trial of self-acupressure to manage the symptom cluster of insomnia, depression, and anxiety in cancer patients undergoing chemotherapy. Sleep Breath. 2022 Mar;26(1):445-456. doi: 10.1007/s11325-021-02370-8. Epub 2021 Apr 14. PMID 33855642

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03823456/Prot_SAP_ICF_000.pdf